CLINICAL TRIAL: NCT03196219
Title: A Phase 2, Open-label and Single-Blind Study to Evaluate the Microbiology, Safety and Tolerability of C16G2 Varnish and Strip Administered in Multiple Doses to Adolescent and Adult Dental Subjects
Brief Title: A Phase 2 Study to Evaluate the Microbiology, Safety and Tolerability of C16G2 Varnish and Strip in Adolescent and Adult Subjects
Acronym: C3J17-206-00
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armata Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: C3J17-206-00
Record Dates: First submitted 2017-06-21; First posted 2017-06-22 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Antimicrobial Peptides

STUDY DESIGN:
Intervention Model Description: Study Arms 1 and 2 will be enrolled in parallel followed by Study Arm 3.
Who Masked: Participant
Masking Description: In the single-blind Study Arm 2, active and placebo will be identical in appearance and labeled in a blinded fashion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: Open-Enrollment Multiple Dose C16G2 Varnish (Experimental): Eight subjects will be enrolled in an open-label manner and will receive a daily dose of C16G2 Varnish application over 3 days followed by 14 doses of C16G2 Strip administered over 7 days. Following the three C16G2 Varnish applications, each subject will receive 7 days of AM and PM dosing with C16G2 Strip.
  Interventions: Drug: C16G2
- Arm 2A: Single-Blind C16G2 Varnish (Experimental): Twelve subjects will be enrolled in a single-blind manner. Subjects will receive four C16G2 Varnish applications over 7 days (Days 0, 2, 5 & 7), followed by 3 additional weekly varnish administrations. The treatment allocation will be 1:1 (6 subjects C16G2 Varnish, 6 subjects Placebo).
  Interventions: Drug: C16G2
- Arm 2B: Single-Blind Placebo (Placebo Comparator): Twelve subjects will be enrolled in a single-blind manner. Subjects will receive Placebo applications over 7 days (Days 0, 2, 5 & 7), followed by 3 additional weekly varnish administrations. The treatment allocation will be 1:1 (6 subjects C16G2 Varnish, 6 subjects Placebo).
  Interventions: Drug: Placebo
- Arm 3: Open-Enrollment Single Dose C16G2 Varnish (Experimental): If initiated, Study Arm 3 will enroll 6 subjects in an open-label manner. Subjects will receive daily single doses of C16G2 Varnish over 10 days, for a total of 10 doses.
  Interventions: Drug: C16G2

INTERVENTIONS:
Drug: C16G2 — C16G2
  Other Names: Antimicrobial Peptide
  Arms: Arm 1: Open-Enrollment Multiple Dose C16G2 Varnish; Arm 2A: Single-Blind C16G2 Varnish; Arm 3: Open-Enrollment Single Dose C16G2 Varnish
Drug: Placebo — Varnish Placebo
  Arms: Arm 2B: Single-Blind Placebo

SUMMARY:
An open-label and single-blind phase 2 study to evaluate the oral microbiology, safety and tolerability of multiple C16G2 Varnish and Strip applications in male and female dental subjects 12-75 years of age. The study will compare multiple study drug administrations of C16G2 Varnish and/or C16G2 Strip in three study arms.

In Study Arm 1 eight subjects will be enrolled in an open-label manner and will receive a daily dose of C16G2 Varnish application over 3 days followed by 14 doses of C16G2 Strip administered over 7 days. Following the three C16G2 Varnish applications, each subject will receive 7 days of AM and PM dosing with C16G2 Strip and will be followed for microbiology for up to 2 months after the last study drug administration.

Study Arm 2 will enroll 12 subjects in a single-blind manner. Subjects will receive four C16G2 Varnish or Placebo applications over 7 days, followed by 3 additional weekly varnish administrations. Subjects will be followed for microbiology for up to 2 months after the last study drug administration.The treatment allocation will be 1:1 (6 subjects receiving C16G2 Varnish, 6 subjects receiving Placebo).

Study Arm 3 will be initiated based on the Sponsor's review of all microbiology data up to two week post last study drug administration from Study Arm 2. If initiated, Study Arm 3 will enroll 6 subjects in an open-label manner. Subjects will receive daily single doses of C16G2 Varnish over 10 days, for a total of 10 doses and will be followed for microbiology for up to 2 months after the last study drug administration.

DETAILED DESCRIPTION:
An open-label and single-blind phase 2 study to evaluate the oral microbiology, safety and tolerability of multiple C16G2 Varnish and Strip applications in male and female dental subjects 12-75 years of age.

The study will compare multiple study drug administrations of 13.6 milligrams (mg) of C16G2 Varnish and 9.2 mg of C16G2 Strip in three study arms. Before dosing of study drug, eligible subjects will receive professional dental prophylaxis between Days -7 and -2.

In Study Arm 1 eight subjects will be enrolled in an open-label manner and will receive a daily dose of C16G2 Varnish application over 3 days followed by 14 doses of C16G2 Strip administered over 7 days. C16G2 Varnish will be applied with a small brush typically used in dental varnish administration. Following the three C16G2 Varnish applications, each subject will receive 7 days of AM and PM dosing with C16G2 Strip. To evaluate the durability of S. mutans suppression, study subjects will be followed for microbiology for up to 2 months after the last study drug administration.

Study Arm 2 will enroll 12 subjects in a single-blind manner. Subjects will receive four C16G2 Varnish or Placebo applications over 7 days (Days 0, 2, 5 & 7), followed by 3 additional weekly varnish administrations. The treatment allocation will be 1:1 (6 subjects receiving C16G2 Varnish, 6 subjects receiving Placebo). To evaluate the durability of S. mutans suppression, study subjects will be followed for microbiology for up to 2 months after the last study drug administration.

Study Arm 3 will be initiated based on the Sponsor's review of all microbiology data up to two week post last study drug administration from Study Arm 2.

If initiated, Study Arm 3 will enroll 6 subjects in an open-label manner. Subjects will receive daily single doses of C16G2 Varnish over 10 days, for a total of 10 doses. To evaluate the durability of S. mutans suppression, study subjects will be followed for microbiology for up to 2 months after the last study drug administration.

Clinic visits in Study Arm 1 include Visit 1 (Screening/Days -30 to -1), Visit 2 (Prophylaxis/Day -7 to -2), Eligibility Confirmation, Baseline & First C16G2 Varnish Dosing at Visit 3, Visits 4 & 5 (C16G2 Varnish Administration), Visits 6-19 (AM & PM C16G2 Strip Administration), Follow-up Visits 20 & 21 (Safety and Microbiology) and Follow-up Visits 22-24 (Microbiology only).

Clinic visits in Study Arm 2 include Visit 1 (Screening/Days -30 to -1), Visit 2 (Prophylaxis/Day -7 to -2), Eligibility Confirmation, Baseline & First C16G2 Varnish or Placebo Dosing at Visit 3, Visits 4-9 (C16G2 Varnish or Placebo Administration), Follow-up Visits 10 & 11 (Safety and Microbiology) and Follow-up Visits 12-14 (Microbiology only).

Clinic visits in Study Arm 3 include Clinic Visit 1 (Screening/Days -30 to -1), Visit 2 (Prophylaxis/Day -7 to -2), Eligibility Confirmation, Baseline & First C16G2 Varnish Dosing at Visit 3, Visits 4-12 (C16G2 Varnish Administration), Follow-up Visits 13 & 14 (Safety and Microbiology) and Follow-up Visits 15-17 (Microbiology only).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 12-75 years of age
2. Adults subjects provide written informed consent and adolescent subjects give written or verbal assent, as appropriate, and parent(s) or legal guardian(s) give written informed consent
3. Female subjects of childbearing potential must agree to use one of the following forms of contraception from screening through the last study visit: hormonal (oral, implant, or injection) begun >30 days prior to screening; barrier (condom, diaphragm, or cervical cap with spermicide); intrauterine device (IUD). Acceptable contraceptive options may also include abstinence, relationship with a same sex partner or partner who has had a vasectomy at least six (6) months prior to the screening visit
4. Negative urine pregnancy test in all females of childbearing potential (past menarche)
5. Male subjects of sexual activity age: willing to use contraception or abstain from sexual activity beginning with the first exposure to study drug and continuing until discharged from the study due to completion or Early Termination
6. Healthy, as determined by the Investigator (in consultation with the Medical Monitor, as needed), based on medical and dental history, concurrent illnesses, laboratory results, concomitant medications, oral cavity assessment, and targeted physical examination (general, extraoral, head and neck) during Screening.

   Note: Subjects on a stable dose of medication may be eligible for screening and will be assessed by the medical monitor on a case-by-case basis.
7. Have a minimum of 12 bicuspids and molars with a minimum of 8 molars and bicuspids NOT having restorations, crowns or sealants
8. Demonstrated ability to expectorate ≥2 mL of stimulated saliva in 5 minutes
9. Have a salivary S. mutans of 1.0 x 10^5 CFUs/mL or greater at Screening using mitis salivarius-bacitracin (MSB) agar plating
10. Willing to refrain from using non-study dentifrice and other non-study oral care products (oral care rinses, fluoride products, etc.) during the study
11. Willing to postpone elective dental procedures (e.g., dental cleanings) between Screening and final post-treatment visit (End of Study or Early Termination)
12. Willing and able to comply with oral hygiene and diet instructions
13. Able to communicate with the Investigator/study center personnel, understand and comply with the study requirements, and willing to return for protocol-specified visits at the appointed times

Exclusion Criteria:

1. Advanced periodontal disease
2. Active caries lesion(s) within 30 days prior to study drug administration (confirmed by comprehensive caries examination including standard radiographs). Subjects presenting with insipient, non-cavitated lesion(s) are not excluded.

   Note: If radiographs are deemed appropriate for the study and taken within 6 months prior to the Screening visit, these may be used for determining eligibility and are not required to be repeated at Screening
3. Partially erupted teeth where the entire crown is not erupted or an operculum is present
4. Medical condition (e.g., artificial heart valve, history of infective endocarditis, cardiac transplant with valvular dysfunction, congenital heart disease or total joint replacement) for which antibiotics are recommended prior to dental visits and/or procedures
5. Pathologic lesions of the oral cavity (suspicious or confirmed)
6. Full dentures or permanent orthodontic appliances, e.g., braces, buccal or lingual brackets. Note: Partial dentures, removable retainers and night guards are not excluded, provided that they are cleaned regularly throughout the duration of the study
7. Use of systemic antibiotics, topical oral antibiotics, any immunosuppressant therapy, and steroids, beginning 30 days prior to Screening until the end of study participation
8. Medical history indicating the woman is pregnant, breastfeeding/lactating or has a positive urine pregnancy test
9. Participation in a clinical trial or receipt of a non-FDA approved therapy within 30 days prior to study drug administration (depending on the specifics, participation in an observational study is not necessarily excluded)
10. Participation in a previous C16G2 clinical trial having received either C16G2 Strip, C16G2 Varnish or Placebo Varnish
11. Presence of any condition or concurrent illness, which in the opinion of the Investigator, would compromise normal immune function (e.g., diabetes, rheumatoid arthritis, lupus, liver disease, organ transplant, etc.), interfere with the use of study dentifrice and oral care products, or interfere with the ability to comply with study requirements, or jeopardize the safety of the subject or the validity of the study results

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pittaway, DMD, Principal Investigator — Plaza West II Dental Group
Locations (1):
- John F. Pittaway, DMD, Kalispell, Montana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment into Study Arms 1 and 2 was concurrent and based on enrollment logistics.
  Study Arm 3 was to be initiated after a microbiology data review of 2-week follow-up data from Study Arm 2. Study Arm 3 was not initiated.
Groups:
- Arm 2A: Single-Blind C16G2 Varnish; Arm 2B: Single-Blind Placebo: Twelve subjects will be enrolled in a single-blind manner. Subjects will receive four C16G2 Varnish or Placebo applications over 7 days (Days 0, 2, 5 & 7), followed by 3 additional weekly varnish administrations. The treatment allocation will be 1:1 (6 subjects C16G2 Varnish, 6 subjects Placebo).
Period: Overall Study
Arm/Group | Arm 1: Open-Enrollment Multiple Dose C16G2 Varnish | Arm 2A: Single-Blind C16G2 Varnish | Arm 2B: Single-Blind Placebo | Arm 3: Open-Enrollment Single Dose C16G2 Varnish
Started | 8 | 6 | 6 | 0
Completed | 8 | 6 | 6 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrollment into Study Arms 1 and 2 was concurrent and based on enrollment logistics.
Groups:
- Arm 2A: Single-Blind C16G2 Varnish; Arm 2B: Single-Blind Placebo: Twelve subjects will be enrolled in a single-blind manner. Subjects will receive four C16G2 Varnish or Placebo applications over 7 days (Days 0, 2, 5 & 7), followed by 3 additional weekly varnish administrations. The treatment allocation will be 1:1 (6 subjects C16G2 Varnish, 6 subjects Placebo).
  C16G2: C16G2
  Placebo: Varnish Placebo
- Total: Total of all reporting groups
Arm/Group | Arm 1: Open-Enrollment Multiple Dose C16G2 Varnish | Arm 2A: Single-Blind C16G2 Varnish | Arm 2B: Single-Blind Placebo | Total
Number analyzed (Participants) | 8 | 6 | 6 | 20
Age, Continuous [Mean (Full Range); unit: years] | 18.8 [12 to 33] | 24.1 [12 to 37] | 24.1 [12 to 37] | 22 [12 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 6 | 4 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 5 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 6 | 20
S. mutans of 1.0 x 105 CFUs/mL or greater [Count of Participants; unit: Participants] | 8 | 6 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Antimicrobial Activity of C16G2
Description: To assess the targeted antimicrobial activity of C16G2 applications as measured by a reduction in Streptococcus mutans in saliva and dental plaque using S. mutans CFUs using mitis-salivarius bacitrain (MSB) agar plating. Streptococcus species present in the oral cavity have been traditionally isolated from oral cavity samples using MSB agar plates. The antimicrobial activity of crystal violet dye, high sucrose content, sodium tellurite and bacitracin effectively prevent the growth of all bacteria except for streptococci. Further differentiation of streptococci is accomplished by observing colony morphology. S. mutans grows in large blue colonies with dry frosted tops or pale blue gumdrops and can be differentiated from other bacterial colonies.
Time Frame: Evaluated over up to 2 months
Population: Enrollment into Study Arms 1 and 2 was concurrent and based on enrollment logistics.
  Study Arm 3 was to be initiated after a microbiology data review of 2-week follow-up data from Study Arm 2. Study Arm 3 was not initiated.
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Arm 1: Open-Enrollment Multiple Dose C16G2 Varnish | Arm 2A: Single-Blind C16G2 Varnish | Arm 2B: Single-Blind Placebo
Number analyzed (Participants) | 8 | 6 | 6
CFU/mL
  Saliva Sample: S. mutans Change from Baseline | -0.49 (0.48) | 0.23 (0.56) | -0.44 (0.51)
  Dental Plaque Sample: S. mutans Change from Baseline | -0.31 (0.38) | -0.22 (0.95) | -0.31 (0.73)

2. Primary Outcome: Total Oral Bacterial Levels
Description: To assess total bacteria in saliva and dental plaque post study drug administration using total bacteria CFUs using Todd Hewitt (TH) agar plating and the log transformed changes from baseline Total Bacteria levels in dental plaque and saliva including N, mean, SD, median and range at each assessment time point following the first administration of C16G2.
Time Frame: 1 day post last study drug administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Arm 1: Open-Enrollment Multiple Dose C16G2 Varnish | Arm 2A: Single-Blind C16G2 Varnish | Arm 2B: Single-Blind Placebo
Number analyzed (Participants) | 8 | 6 | 6
CFU/mL
  Saliva Sample - Total Bacteria by TH Agar Plating from Baseline | 0.001 (0.24) | 0.075 (0.28) | -0.155 (0.130)
  Dental Plaque Sample - Total Bacteria by TH Agar Plating from Baseline | -0.214 (0.312) | -0.21 (0.63) | -0.18 (0.42)

3. Secondary Outcome: To Evaluate the Safety of Multiple C16G2
Description: Safety will be assessed by performing targeted physical examinations, oral cavity exams, taking vital signs and collection of adverse events categorized according to system organ class (SOC) and preferred term (PT) based on coding to the Medical Dictionary for Regulatory Activities (MedDRA®), Version 17.1. Comprehensive examinations of oral hard and soft tissue structures, as well as targeted exams of specific musculoskeletal and extraoral sites were performed at selected time points; vital signs (blood pressure, heart rate and temperature) were taken.
Time Frame: Up to 7 days post last study drug administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Open-Enrollment Multiple Dose C16G2 Varnish | Arm 2A: Single-Blind C16G2 Varnish | Arm 2B: Single-Blind Placebo
Number analyzed (Participants) | 8 | 6 | 6
Participants
  Participants with Adverse Events Related to Study Drug | 0 | 0 | 0
  Participants with Clinical Significant Oral Cavity Changes | 0 | 0 | 0
  Participants with Clinical Significant Vital Sign Changes | 0 | 0 | 0
  Participants with Abnormal Physical Exam Findings | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 months
Description: Enrollment into Study Arms 1 and 2 was concurrent and based on enrollment logistics.
  Study Arm 3 was to be initiated after a microbiology data review of 2-week follow-up data from Study Arm 2. Study Arm 3 was not initiated.
  Arm 3: Not enrolled. Therefore number of particpants at risk for Serious Adverse Events, All-Cause Mortality, and other (Not Including Serious) Adverse Events is zero.
Arm/Group | Arm 1: Open-Enrollment Multiple Dose C16G2 Varnish | Arm 2A: Single-Blind C16G2 Varnish | Arm 2B: Single-Blind Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03196219/Prot_SAP_000.pdf